CLINICAL TRIAL: NCT05675124
Title: Prospective Randomized Comparison of Needlescopic Versus Conventional Laparoscopic Adrenalectomy for Unilateral Adrenal Tumors Less Than 4 cm in Diameter Among Patients With Primary Aldosteronism
Brief Title: Comparison of Needlescopic vs. Conventional Laparoscopic Adrenalectomy for Tumor Less Than 4 cm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 202204074RINC
Record Dates: First submitted 2022-08-19; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Post Operative Pain, Acute
Keywords: Visual Analogue Scale; Post Operative Pain; Dosage of analgesic; Cosmetic
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needlescopic laparoscopic adrenalectomy (Experimental): Needlescopic laparoscopic surgery refers to the use of instruments with a diameter of less than or equal to 3 mm for laparoscopic surgery.
  Interventions: Device: Needlescopic laparoscopic adrenalectomy
- conventional laparoscopic adrenalectomy (Active Comparator): a 12 mm camera port ,and two additional (left anterior axillary line and left midclavicular line; for left tumors) or three additional(right anterior axillary line, right midclavicular line, and subxiphoid; for right tumors) 5 mm working ports along the ipsilateral subcostal were created regionally.
  Interventions: Device: conventional laparoscopic adrenalectomy

INTERVENTIONS:
Device: Needlescopic laparoscopic adrenalectomy — Compared with traditional laparoscopic surgery using 5-12 mm instruments, the wound of needlescopic laparoscopic surgery is smaller. Postoperative pain and recovery are also better than traditional laparoscopic surgery.
  Arms: Needlescopic laparoscopic adrenalectomy
Device: conventional laparoscopic adrenalectomy — conventional laparoscopic adrenalectomy
  Arms: conventional laparoscopic adrenalectomy

SUMMARY:
The investigator conduct a randomized clinical trial for the needlescopic and conventional laparoscopic adrenalectomy to assess whether mini laparoscopic adrenalectomy is better than conventional laparoscopic adrenalectomy in terms of pain, complication rate , and wound cosmetics

DETAILED DESCRIPTION:
If the participant with unilateral PA tumor less than 4cm is willing to enter the clinical trial, he/she will be randomly assigned to two groups (conventional vs needlescopic laparoscopic adrenalectomy) in a 1:1 ratio, followed by preoperative assessement. All procedures were performed by experienced laparoscopic urologists (number of complex laparoscopic procedures > 50 cases/yr for 10 yrs). The participant were blinded to the type of surgical procedure underwent until the pain assessment was completed in the morning of the second days after surgery

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 20 years old.
2. Primary aldosteronism with unilateral adrenal lesions smaller than 4 cm
3. Indications for laparoscopic surgery.
4. Informed consent

Exclusion Criteria:

1. Over 80 years old
2. Suspected adrenal malignancy or pheochromocytoma
3. Other concurrent surgery
4. Patients who underwent bilateral adrenal tumor resection at the same time
5. History of peritonitis or having undergoing major ipsilateral abdominal surgery.
6. American Society of Anesthesiologists (ASA) Class III or IV (with severe cardiovascular disease, uncontrolled hypertension, diabetes, chronic pulmonary obstructive pulmonary disease, morbid obesity (BMI > 40), dialysis patients, myocardial infarction, stroke, coronary artery disease, liver or coagulation dysfunction, etc.)
7. Opioid addiction
8. Patient have side effects from taking of acetaminophen, celecoxib or opioids
9. Acute intoxication of alcohol, sleep aids, anesthetics, centrally acting analgesics, opium or psychotropic drugs has occurred.
10. Patients using monoamine oxidase inhibitors (MAOIs) concurrently or within the past 14 days.
11. Patients with chronic pain or respiratory depression (such as chronic obstructive pulmonary disease)
12. Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Timing that two consecutive VAS less than 3 points | up to 1 month postoperatively
  Timing that two consecutive VAS less than 3 points after operation
  * The nurse for pain assessement would not know the allocation of the patient to this trial arms
  * Wound pain was assessed on a visual analogue scale (VAS) from 0 (none) to 10 (worst)

SECONDARY OUTCOMES:
Cumulative morphine dosing | Right after adrenalectomy until the morning of post-op Day 2 ( before the wound dressing change)
  >On the operative day: morphine (10mg/1mL/amp) 2mg IV Q4H PRN(every 4 hours.Pro re nata) was administered intravenously.
  > Post-op Day 1: acetaminophen (500mg/tab) # 1 PO QID (quater in die) and celecoxib (200 mg/Cap) # 1 PO QD( quaque die), morphine (10mg/1mL/amp) 2mg IV Q4H PRN (every 4 hours.Pro re nata) as rescue analgesia (as VAS >=3)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Chueh, Principal Investigator — Dep. of Urology, NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao CH, Lai MK, Li HY, Chen SC, Chueh SC. Laparoscopic adrenalectomy using needlescopic instruments for adrenal tumors less than 5cm in 112 cases. Eur Urol. 2008 Sep;54(3):640-6. doi: 10.1016/j.eururo.2007.12.028. Epub 2007 Dec 26. PMID 18164803
- [Background] Chueh SC, Chen J, Chen SC, Liao CH, Lai MK. Clipless laparoscopic adrenalectomy with needlescopic instruments. J Urol. 2002 Jan;167(1):39-42; discussion 42-3. doi: 10.1016/s0022-5347(05)65378-5. PMID 11743271